CLINICAL TRIAL: NCT03353935
Title: Functional Outcomes of Nerve-sparing Laparoscopic Eradication of Deep Infiltrating Endometriosis: a Prospective Analysis Using Validated Questionnaires
Brief Title: Functional Outcomes After Nerve Sparing Surgery for Deep Endometriosis
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Stefano Uccella, Doctor, Università degli Studi dell'Insubria
Other Study IDs: 630
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Endometriosis
Keywords: surgery; pelvic function
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NERVE SPARING: Patients who underwent surgery for deep endometriosis were submitted to surgical procedures aiming at sparing the pelvic ortho- and parasympathetic nerves. The subjects were then followed with interviews using validated questionnaires, to assess the possible changes in post-operative urinary sexual and fecal function.
  Interventions: Other: Validated questionnaires

INTERVENTIONS:
Other: Validated questionnaires — Patients were administered pre- and post-operatively the three validated questionnaires ((FSFI, ICIQ-UI short form Italian, NBD score) investigating sexual, urinary, and fecal function, respectively.

SUMMARY:
Patients who underwent surgery for deep endometriosis were submitted to procedures aiming at sparing the pelvic autonomic nervous system. They were observed prospectively followed and interviewed in order to evaluate functional outcomes after surgery.

DETAILED DESCRIPTION:
Surgical tretament for deep endometriosis can produce lesions at the level of the pelvic autonomic system.

Before surgery and 3-12 months after the nerve-sparing surgical procedures, patients were assessed for urinary, sexual and fecal function, in order to evaluate whether sparing of the nerves during the intervention had a beneficial impact on post-operative pelvic function.

ELIGIBILITY:
Inclusion Criteria:

* Deep endometriosis
* Surgical treatment
* Single surgeon

Exclusion Criteria:

* Lost to follow-up
* unwillingness to answer the interview

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients undergoimg nerve-sparing surgery for deep endometriosis were enrolled if they were operated by a single surgeon with extensive background in minimally-invasive pelvic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Pelvic function | 6-12 months
  Any change in urinary, sexual or fecal function after surgery, compared to pre-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Uccella, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- Department of Obstetrics and Gynecology Universita' Dell'Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: No